CLINICAL TRIAL: NCT06317389
Title: PACOME (PAtient Cancer Oral MEdication) Cohort of Patients Treated With Oral Anticancer Drugs Benefiting From Oncoral Multidisciplinary Monitoring in Real Life: Predictive Factors and Safety of Treatments
Acronym: PACOME
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1237
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Oncology; Oncoral Program
Keywords: Cancer outpatient; Oral anticancer drugs; Oncoral; Real-life
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncoral patients: All adult patients with cancer, treated with oral anticancer drugs and benefiting of the ONCORAL program at the Lyon-Sud hospital
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Patients will benefit of supervision by the ONCORAL team in the usual way and their intervention will be limited to completing questionnaires.

SUMMARY:
With the shift to ambulatory care and the rise of ATCO oral anticancer drugs, a growing number of cancer patients are benefiting from oral treatment in an outpatient setting, which meets their needs and preference over injectable chemotherapy with more autonomy and less time spent in the hospital. However, outside the safe hospital context, the complex pharmacological profile of ATCO exposes patients to iatrogenic drug risks. These medicinal problems or Drug Related Problems DRP linked to ATCO are sources of dosage modifications and lead to sub-therapeutic doses compared to clinical trials and consequently to a reduction, in life actual, dose-intensity and expected response. Furthermore, insufficiently controlled in an ambulatory environment and due to a lack of city-hospital coordination, DRPs lead to an increase in the consumption of care.

Oncoral is the pioneering multidisciplinary city-hospital monitoring of outpatients treated with oral anticancer drugs. Set up in 2014 by the Hospices Civils de Lyon, this educational monitoring is based on a tripartite hospital intervention (oncologist, pharmacist, nurse) and a structured city-hospital link with private health professionals (attending doctor, community pharmacist and freelance nurse). Multidisciplinary interventions are focused on PROs and DRPs and combine an educational approach for the patient based on their needs and potential social vulnerabilities.

The PACOME real-life database will describe the population of ambulatory patients treated by ATCO benefiting from the secure multidisciplinary city-hospital Oncoral pathway with the aim of improving knowledge on this population, on the real-life use of ATCO and on new methods of organizing ambulatory cancer care.

The PACOME database collects sociodemographic, clinical and therapeutic data, and experiences in this population. Patients quality of life and other PROs (symptoms and adverse effects experienced by patients), social determinants, health care consumption, the caregiver-patient relationship, the use of digital technology in health, the organization of care, the city-hospital link (interventions of actors and their temporality).

This base will make it possible to optimize the treatment of patients at the individual and population level and to generate evidence in addition to clinical trials, which are expected by health professionals and decision-makers. With patient data from the secure Oncoral pathway, PACOME brings together the three major and inseparable assets of real-life databases: quality, completeness and meaning of the data. It constitutes a basis for essential academic and private collaborations for studies on data and comparative observational or interventional studies, which will contribute to the animation of the new ecosystem of real-life health data in oncology.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18
* eligible for treatment with oral anticancer drug (ATCO) (excluding clinical trial) in a cancer indication and whose treatment with an oral anticancer drug is scheduled
* follow-up in one of the following departments at Lyon-Sud hospital: pulmonology, dermatology, hematology, medical oncology, gastroenterology or radiotherapy.
* without a major psychiatric disorder likely to hinder the progress of the study, in the opinion of the investigator
* participant in the ONCORAL monitoring program
* Not having opposed participating in the study

Exclusion Criteria:

* in an institution
* under legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients eligible for treatment with oral anticancer drugs (excluding clinical trials), followed at Lyon-Sud Hospital and benefiting from the ONCORAL programme.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Relative-Dose-Intensity (RDI) in real life with a prospective follow-up of 6 months within the limit of the duration of treatment with oral anticancer drugs by setting up a data platform for adult patients taking oral anticancer drugs | 1, 3 and 6 months
  Value of RDI (Relative-Dose-Intensity) is the ratio between the dose prescribed to the patient versus the maximum reference dose recommended by the product characteristics summary of the drug.
  This ratio is expressed as a percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Sud - Unité de Pharmacie Clinique Oncologique, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: Undecided